CLINICAL TRIAL: NCT00821275
Title: Multi-Center Clinical Trial of Uterine Artery Embolization Treatment of Uterine Leiomyoma
Brief Title: Clinical Trial of Uterine Artery Embolization for Uterine Leiomyoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Hong Shan, the third Affiliated Hospital of Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007026
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Leiomyoma
Keywords: Uterine Artery Embolization; Leiomyoma; myomectomy; hysterectomy; pregnancy; complication; ovarian function; quality of life
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pregnancy expectation (Active Comparator): The patients who desire for future pregnancy will enroll into this arm , and will be divided into UAE group and SURGERY group.
  Interventions: Procedure: Interventional radiological or surgical management
- No pregnancy expectation (Active Comparator): The patients who don't desire for reserving uterus and/ or future pregnancy will enroll into this arm , and will be divided into UAE group and SURGERY group.
  Interventions: Procedure: Interventional radiological or surgical management

INTERVENTIONS:
Procedure: Interventional radiological or surgical management — Uterine artery embolization will be done for the patients who enroll into UAE group and desire for future pregancy and reserving uterus.Myomectomy will be performed for the patients who enroll into SURGERY group and desire for future pregancy and reserving uterus.Hysterectomy will be done for the patients who enroll into SURGERY group and don't desire for reserving uterus and/or future pregnancy.

SUMMARY:
The efficacy and safety of uterine artery embolization, as compared with standard surgical methods, for the treatment of symptomatic uterine fibroids remain uncertain. The purpose of this trial is to evaluate the uterine volume and tumor size reduction, symptomatic relief, complication, fertility, ovarian function and quality of life with uterine artery embolization for uterine fibroids comparing with standard surgical methods.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of symptomatic uterine leiomyoma

Exclusion Criteria:

* pregnancy
* iodine agent allergy
* patient refuse to take part in this trial
* tumour size is less than 3cm or beyond 10cm
* with endometriosis
* with malignant diseases
* with abnormal coagulation function which can't restore
* with acute inflammatory diseases or acute episode of chronic inflammatory diseases
* with severe heart, lung, liver and kidney, et al. organ diseases.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900 (Estimated)
Dates: Start 2008-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
quality of life | 1,3,5,10 year.
pregnant | 3 years

SECONDARY OUTCOMES:
tumor recurrence | 1,3,5,10 years
complications | 3,6,12,24 months
ovarian functions | 3,6,12 months, 2,3,5 and 10 years
symptom relief | 3,6,12,24 months
tumour volume | 3,6,12 18 24 months and 3,5,10 years

CONTACTS AND LOCATIONS:
Overall Officials: Hong Shan, M.D., PHD., Study Director — Third Affiliated Hospital, Sun Yat-Sen University
Locations (4):
- China (4):
  - Nanfang Hospital of Nanfang medical University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - the first Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University, Guangzhou, Guangdong

REFERENCES:
- See also: The Third Affiliated Hospital of Sun Yat-sen University — http://www.zssy.com.cn/